CLINICAL TRIAL: NCT05281705
Title: Feasibility@ 48: A Cross Sectional Multi-centre Study of Intensive Care Unit (ICU) Mobility Practices Across the United Kingdom.
Brief Title: Feasibility@48: Cross Sectional Study of Intensive Care Unit Mobility Practices Across the United Kingdom
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE:125652 IRAS:262426
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness; Rehabilitation
Keywords: Physiotherapy; Rehabilitation; Mobilisation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intensive Care Unit (ICU) patients commonly experience muscle loss at a rate of 2-3% day. Traditionally, critically ill patients have been managed in bed, however current research suggests that prolonged bedrest cause mechanical silencing of the muscles and exacerbates this muscle wasting. This ICU acquired weakness (ICUAW) leads to poor functional outcome and higher mortality. Research suggests that early out-of-bed mobilisation should occur within 48-hours of ICU admission to militate against this risk, however, this is only achieved in 30% of cases. Common barriers to mobilisation are unstable blood pressure, ventilation, sedation and fatigue. It is plausible that 48-hours is an unrealistic timeframe for mobilisation.

The aim of this study is to explore the mobility practices on a given day in UK adult ICUs. The objectives are to:

1. Determine the level of mobility that is achieved by each patient on adult ICUs, on a given day in the UK.
2. Determine the typical physiological profile of patients on ICU that are both able and unable to participate in antigravity exercise
3. Determine the proportion of adult ICU admissions that achieve out of bed mobilisation in the first 48-72 hours
4. Explore clinician decision making about mobilisation

This is a multi-centre cross-sectional study on one-day only. Over a 24-hour period data will be collected for all ICU patients at the participating centres. The lead physiotherapist will record the highest level of mobility achieved that day, and the physiological parameters from clinical observations. The reasons for the level of mobility achieved will be ranked in order of importance. These data are routinely collected. Data will be anonymised.

Data will be analysed to determine feasibility of mobilisation at 48hours and develop a flow diagram of mobilisation decision-making.

ELIGIBILITY:
Inclusion Criteria:

All patients who are admitted to a participating ICU on the study day will be included

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient in level 2 & 3 ICU beds in the UK
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving a ICU mobility scale more than 3 on the day of the study | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Black C, Sanger H, Battle C, Eden A, Corner E. Feasibility of mobilisation in ICU: a multi-centre point prevalence study of mobility practices in the UK. Crit Care. 2023 Jun 1;27(1):217. doi: 10.1186/s13054-023-04508-4. PMID 37264471